CLINICAL TRIAL: NCT00048022
Title: Inhaled Corticosteroid Replacement Study - Efficacy and Safety of Ro 27-2441 (Test Drug) in Moderate Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: BA16630
Record Dates: First submitted 2002-10-24; First posted 2002-10-25 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: Dual Integrin Antagonist

SUMMARY:
The primary objective of the study is to evaluate the anti-inflammatory action and safety of Ro 27-2441 (study drug) in asthmatic patients currently taking inhaled corticosteroids. The research is being conducted at up to 40 clinical research sites in the US. Study participants will have a number of visits to a research site over a 4-month period.

ELIGIBILITY:
Inclusion Criteria:

* Persistent asthma for more than 1 year
* Currently receiving treatment with a stable dose of inhaled corticosteroids for more than 3 months
* In good health as demonstrated by medical history and physical exam
* Negative urine pregnancy test
* Commitment to use two forms of effective contraception simultaneously throughout the study duration and for 1 month after discontinuing therapy

Exclusion Criteria:

* Hospitalization for treatment of asthma and/or treatment with oral/injectable corticosteroids within 3 months before the start of the study
* Undergoing allergy shots unless on a stable maintenance dose for 3 months before the start of the study
* History of chronic pulmonary diseases other than asthma
* Treatment of conditions other than asthma with oral corticosteroids within 1 month of the start of the study
* Current tobacco usage
* Smoking history of greater than 10 pack-year history of cigarette smoking (number of packs smoked per day times the number of years smoked)
* History or evidence of drug or alcohol abuse
* Diagnosis or evidence of an infectious illness within one month of Visit 1
* Clinically significant diseases as assessed by the study doctor
* Participation in another clinical study with an experimental drug within one month of start of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10-25 (Actual); Primary Completion 2004-02-02 (Actual); Study Completion 2004-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (53):
  - Huntington Beach, California
  - Los Angeles, California
  - Mission Viejo, California
  - San Diego, California
  - San Jose, California
  - Walnut Creek, California
  - Boulder, Colorado
  - Denver, Colorado
  - Louisville, Colorado
  - Sarasota, Florida
  - Tallahassee, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Normal, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Lenexa, Kansas
  - Metairie, Louisiana
  - North Dartmouth, Massachusetts
  - Ypsilanti, Michigan
  - Missoula, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Forked River, New Jersey
  - Teaneck, New Jersey
  - Farmingdale, New York
  - Rochester, New York
  - Rockville Centre, New York
  - Asheville, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Medford, Oregon
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Upland, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Sugar Land, Texas
  - Murray, Utah
  - South Burlington, Vermont
  - Abingdon, Virginia
  - Bellingham, Washington
  - Kirkland, Washington
  - Seattle, Washington
  - Tacoma, Washington
  - Morgantown, West Virginia
  - Madison, Wisconsin
- Ponce, Puerto Rico